CLINICAL TRIAL: NCT04750863
Title: Evaluation of Adult Onset Still Disease Classification Criteria and Differential Diagnosis at Eighteen Months of Follow-up
Acronym: AOSD-DIF
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2021PI001
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Adult Onset Still Disease
Keywords: adult onset still disease; differential diagnosis; diagnosis performance
MeSH Terms: conditions — Still's Disease, Adult-Onset

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: diagnosis criteria performance

SUMMARY:
Adult Onset Still Disease (AOSD) is an acquired inflammatory disease of unknown etiology, presenting with non specific symptoms. Its diagnosis rely on sets of criteria, i.e. Fautrel Criteria and Yamaguchi Criteria. However, differential diagnosis might appear during follow-up of patients. The aim of this study is to assess diagnostic performance of Fautral and Yamaguchi Criteria after 18 months of follow-up, and to describe differential diagnosis appearing during follow-up.

DETAILED DESCRIPTION:
Adult Onset Still Disease (AOSD) is an acquired inflammatory disease of unknown etiology, presenting with non specific symptoms. Other conditions such as cancer, infection or other inflammatory disease might mimick its symptoms. Its diagnosis rely on sets of criteria, i.e. Fautrel Criteria and Yamaguchi Criteria. However, differential diagnosis might appear during follow-up after an initial diagnosis of AOSD. The aim of this study is to assess diagnostic performance of Fautral and Yamaguchi Criteria after 18 months of follow-up, and to describe differential diagnosis appearing during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* adults
* with glycosylated ferritin dosage for suspected adult onset still disease
* with at least 18 month of follow-up

Exclusion Criteria:

* known infectious disease
* known cancer
* known active connective tissue disease or vasculitis

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with suspected adult onset still disease with at least 18 months of follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2010-07-15 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
diagnosis performance of Yamaguchi and Fautrel criteria at 18 months of follow-up | after 18 months of follow-up
  Sensitivity, Specificity, positive predictive value, negative predictive value

SECONDARY OUTCOMES:
description of differential diagnosis mimicking adult onset still disease | after 18 months of follow-up
identifying factors associated with the occurence of a differential diagnosis during follow-up | after 18 months of follow-up

IPD SHARING:
Plan to Share IPD: No